CLINICAL TRIAL: NCT06362369
Title: A Phase 1b/2a Multi-Center, Dose Escalation and Reference Regimen-Controlled, Multi-Cohort Study to Determine the Safety and Efficacy of Oral 7HP349 (Alintegimod) in Combination With Ipilimumab Followed by Nivolumab Monotherapy in Patients With Locally Advanced or Metastatic Cancers Following One or More Prior Therapies
Brief Title: A Study of Oral 7HP349 (Alintegimod) in Combination With Ipilimumab Followed by Nivolumab Monotherapy
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: 7 Hills Pharma, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 7HP-111
Record Dates: First submitted 2024-03-21; First posted 2024-04-12 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Advanced Cancer; Advanced Solid Tumor; Melanoma; Metastasis; Pleural Mesothelioma; Renal Cell Carcinoma; MSI-High; Mismatch Repair Deficiency; Colorectal Cancer; Hepatocellular Carcinoma; Hepatocellular Cancer; Renal Cell Cancer; Kidney Cancer; Skin Cancer; Non Small Cell Lung Cancer; NSCLC; Anaplastic Lymphoma Kinase Genomic Tumor Aberrations; ALK Genomic Tumor Aberrations
Keywords: Phase 1; Phase 1b; 7 Hills Pharma
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis; Mesothelioma, Malignant; Carcinoma, Renal Cell; Turcot syndrome; Colorectal Neoplasms; Carcinoma, Hepatocellular; Liver Neoplasms; Kidney Neoplasms; Skin Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Ipilimumab; Nivolumab

STUDY DESIGN:
Masking Description: Phase 1b - Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dose Escalation - Open Label Phase 1b (Experimental): Alintegimod dose escalation, 4 cohorts Alintegimod monotherapy 1 cycle Alintegimod + Ipilimumab - 4 cycles Nivolumab - 11 cycles
  Interventions: Drug: Alintegimod; Drug: Ipilimumab; Drug: Nivolumab

INTERVENTIONS:
Drug: Alintegimod — Alintegimod will be provided in bottles of 30 softgel capsules for oral administration
  Other Names: 7HP349
Drug: Ipilimumab — Ipilimumab (Yervoy) will be administered via IV
  Other Names: Yervoy
Drug: Nivolumab — Nivolumab (Opdivo) will be administered via IV
  Other Names: Opdivo

SUMMARY:
This study is an open-label Phase Ib (Part A) dose escalation followed by a blinded, randomized, multi cohort Phase 2a (Part B) comparison of combination vs. reference regimens.

Currently study will only be enrolling the Phase 1b and the Phase 2a protocol requirements will be added to the study near completion of the Phase 1b

DETAILED DESCRIPTION:
This Phase study is designed to evaluate the safety, tolerability, and preliminary efficacy of oral Alintegimod (Alintegimod) alone, and then in combination with ipilimumab for, followed by nivolumab monotherapy cycles. All patients will receive nivolumab after completion of treatment with Alintegimod plus ipilimumab combination therapy to continue nivolumab treatment until the end of study (12 months) unless progression or toxicity result in early termination.

ELIGIBILITY:
Inclusion and Exclusion Criteria for Phase 1b

Inclusion Criteria

1. Adult patients (age 18 or older)
2. Patient has a histologically confirmed diagnosis of any of the following locally advanced or metastatic solid tumors: melanoma, pleural mesothelioma, renal cell carcinoma, MSI-high or mismatch repair-deficient colorectal cancer, hepatocellular carcinoma, and non-small cell lung cancer with no EGFR or anaplastic lymphoma kinase (ALK) genomic tumor aberrations, or tumor types for which the combination of ipilimumab and nivolumab has been FDA approved. Patients may have received treatment with anti PD-1/PD-L1.
3. ANC ≥ 1000/µL without use of G-CSF, Hgb ≥ 9 g/dL without required blood transfusion for at least 5 days prior to pretreatment baseline, and platelet count ≥ 75,000/µL without transfusions for at least 5 days prior to pretreatment baseline.
4. ECOG performance status of 0 or 1.
5. Has a life expectancy of > 12 weeks.
6. Renal and hepatic function requirements:

   * a. Renal function with either an eCrCL ≥ 60 mL/min (modified Cockcroft-Gault) or eGFR ≥ 60 mL/min/1.73 m2 (using MDRD or CKD-EPI or similar equations).
   * b. Hepatic function with ALT/AST ≤ 3 x ULN, total bilirubin ≤ 1.5 x ULN (except for patients with Gilbert Syndrome). If patients have hepatic metastases, then AST/ALT≤ 5 x ULN will be allowed.
7. Men receiving the investigational drug and are sexually active with women of child-bearing potential (WCBP) must use contraception during treatment and for 5 half-lives after the last dose of the investigational drug or Women, not otherwise meeting other exclusion criteria, who are WCBP must be on contraception for a minimum duration of 3 months prior to treatment and continue contraception during treatment and for 5 half-lives after the last dose of the investigational drug.
8. All Grade 3 AEs related to prior therapies have returned to Grade 1 or resolved to baseline (this includes with appropriate therapy in the case of thyroid dysfunction).
9. All patients must have measurable disease by applicable RECIST criteria.
10. Willing to allow blood samples to be used for research.

Exclusion Criteria:

1. Patients must not have received prior anticancer therapy or radiation therapy within the 3 weeks and must not have undergone major surgery within 4 weeks prior to initiation of treatment on protocol. Palliative radiation therapy is allowed. For small molecules (MW < 0.9 kDA), the washout period is 3 weeks or 5 half-lives, whatever comes first.
2. Active brain metastasis or leptomeningeal disease. Patients with treated brain metastasis must have stable disease, evidenced by MRI brain imaging for at least 4 weeks, and the patient must have been off steroids for at least 2 weeks prior to first dose of study drug.
3. Previous episodes of ≥ Grade 3 (G3) immune-related toxicity that includes G3 colitis, G3 pneumonitis, G3 skin rash, G3 increase in liver enzymes (with the exception of symptoms that in the opinion of the investigator will not compromise the patients' safety on the trial. Patients with stable endocrinological AEs (e.g., hypothyroidism, adrenal insufficiency, hypopituitarism, or diabetes mellitus) are allowed.
4. Persistent toxicity of NCI CTCAE version 5 Grade > 1 severity that is related to prior therapy.

   Note: Sensory neuropathy, hypothyroidism or alopecia of Grade ≤ 2 are acceptable. Other Grade 2 toxicities of prior treatments that are controlled with medication (e.g., diabetes or hypertension) are permitted.
5. Concurrent administration of medications or foods that are strong inhibitors or inducers of cytochrome p450 3A (CYP3A) within 2 weeks before study intervention. Alintegimod may increase exposure to CYP3A4 substrates; consider a dose reduction of such substrates and monitor for signs of toxicities of co-administered sensitive CYP3A substrates (see listing of strong inhibitors and inducer drugs in FDA tables). An alternative is to replace such agents with drugs that are not CYP3A4 metabolized if at all feasible.
6. The patient has cardiac conditions as follows:

   * a) myocarditis;
   * b) uncontrolled hypertension (blood pressure > 160/100) despite optimal therapy;
   * c) uncontrolled angina; ventricular arrhythmias; congestive heart failure (New York Heart Association Class II or above);
   * d) prior or current cardiomyopathy;
   * e) uncontrolled atrial fibrillation with heart rate > 100 beats per minute (bpm); unstable ischemic heart disease (myocardial infarction within 6 months prior to starting treatment or angina requiring use of nitrates more than once weekly);
   * f) concomitant medication with drugs known to cause Torsades de Pointes;87
   * g) QT interval correction for heart rate using Fridericia's formula (QTcF) ≥ 470 ms (average from 3 QTcF values on the triplicate 12-lead electrocardiogram [ECG]) at screening.
7. Known history of a positive test for HIV, or positive test for hepatitis B (positive for HBsAg) or hepatitis C (HCV RNA).
8. Concurrent malignancies are permitted if they were previously treated, and all treatment of that malignancy was completed at least 2 years before enrollment and no evidence of disease exists, or with agreement from the Principal Investigator (PI), patients who have a concurrent malignancy that is clinically stable and does not require tumor-directed treatment are eligible to participate if the risk of the prior malignancy interfering with either safety or efficacy endpoints is very low, or with agreement from the PI, other malignancies may be permitted if the risk of the prior malignancy interfering with either safety or efficacy end points is very low. Adequately treated basal or squamous cell carcinoma or carcinoma in situ is allowed.
9. Men receiving the investigational drug and are sexually active with women of child-bearing potential (WOCBP) must use contraception during treatment and for 5 half-lives after the last dose of the investigational drug or Women, not otherwise meeting other exclusion criteria, who are WOCBP must be on contraception for a minimum duration of 3 months prior to treatment and continue contraception during treatment and for 5 half-lives after the last dose of the investigational drug.
10. The patient has concurrent severe and/or uncontrolled medical disease that could compromise participation in the study (i.e., uncontrolled diabetes, severe infection requiring active treatment, severe malnutrition, chronic severe liver or renal disease).
11. Use of corticosteroids or other immunosuppressive medication, current or within 14 days of administration of Alintegimod with the following exceptions:

    * a) Topical, intranasal, inhaled, ocular, intra-articular corticosteroids;
    * b) Physiological doses of replacement corticosteroids (e.g., for adrenal insufficiency) are not to exceed 10 mg/day of prednisone or equivalent.
    * c) Corticosteroid premedication for infusion and/or hypersensitivity reactions.
    * d) Patients may be treated with a short (<24h) pulse course of corticosteroids to mitigate infusion or hypersensitivity reactions to radiocontrast agents.
12. Receipt of live attenuated vaccine within 28 days of the first dose of Alintegimod.
13. Serious autoimmune disease at the discretion of the treating Investigator: patients with a history of active serious inflammatory bowel disease (including Crohn's disease and ulcerative colitis) and autoimmune disorders such as rheumatoid arthritis, systemic progressive sclerosis (scleroderma), systemic lupus erythematosus or autoimmune vasculitis (e.g., Wegener's Granulomatosis) are excluded from participation in this study
14. Active or history of pneumonitis (drug-induced), idiopathic pulmonary fibrosis, Interstitial Lung Disease (ILD), or lung disease that may interfere with assessment of pneumonitis. History of radiation pneumonitis in a previous radiation field is permitted.
15. Previous participation in a study of any investigational agent within 21 days of enrollment or within 5 half-lives of the study treatment, whichever is the least.
16. Use of mechanical ventilation or having a resting O2 saturation < 90% (on room air) by pulse-oximetry, require renal dialysis, require vasopressors, and/or severe hepatic sinusoidal obstruction syndrome.
17. Proven or suspected ongoing systemic infection requiring IV antibiotics.
18. Women who are pregnant or lactating.

    Note: Women of childbearing potential (WOCBP) must have a "negative" serum pregnancy test within 1 week prior to treatment. Non-childbearing potential is defined as 1 of the following:
    * a) Postmenopausal with > 1 year since last menses and:
    * 1. If ≥ 65 years old, follicle-stimulating hormone (FSH) > 40 mIU/mL.
    * 2. If ≥ 65 years old and not on hormone replacement therapy (HRT), FSH > 30 mIU/mL.
    * 3. If ≥ 65 years old and on HRT, the FSH requirement is not applicable. Postmenopausal females on HRT will be allowed if HRT has been stable for ≥ 6 months prior to dosing of study drug(s).
    * b) Written medical documentation of being sterilized (e.g., hysterectomy, double oophorectomy, bilateral salpingectomy) with the procedure performed ≥ 6 months prior to dosing study drug(s).

    Note: Tubal ligation is not considered a form of permanent sterilization.
19. Psychiatric illness/social circumstances that would limit compliance with study requirements and substantially increase the risk of adverse events or have compromised ability to provide written informed consent.
20. Patients who have had allogeneic tissue or solid organ transplantation. Prior T cell therapy is allowed
21. Use of biotin (i.e., Vitamin B7) or supplements containing biotin higher than the daily adequate intake of 30 µg (NIH-ODS 2022; Section 5.9.2.1).

    Note: Patients who switch from a high dose to a dose of ≤30 µg/day are eligible for study entry.
22. Any condition that is in the opinion of the investigator may compromise patient's participation in the trial.
23. Active peptic ulcer disease or gastritis, active diverticulitis, or other serious gastrointestinal disease associated with diarrhea within the past 2 years before the start of therapy or GI disease which affects oral drug absorption.
24. Patients with known soy allergy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2024-08-23 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants treated with Alintegimod monotherapy with treatment related adverse events as assessed by CTCAEv5.0 | 1 year
  To evaluate the safety and tolerability of Alintegimod administered as monotherapy, in the patients with adverse events as assessed by CTCAE v5.0 and coded by System Organ Class (SOC) using MedDRA coding dictionary
Number of participants treated with Alintegimod in combination with treatment related adverse events as assessed by CTCAEv5.0 | 1 year
  To evaluate the safety and tolerability of Alintegimod administered in combination with ipilimumab followed by sequential nivolumab monotherapy, in the number of patients with adverse events as assessed by CTCAE v5.0 and coded by System Organ Class (SOC) using MedDRA coding dictionary
Define RPTDs for Alintegimod | 18 months
  To define two doses of the Alintegimod + ipilimumab followed by nivolumab cohorts that will be used in the Phase 2a (Part B) study.

SECONDARY OUTCOMES:
Characterize Pharmacokinetics of Alintegimod monotherapy by measuring Maximum Plasma Concentration (Cmax) | 1 year
  To characterize the pharmacokinetics of Cmax of Alintegimod monotherapy.
Characterize Pharmacokinetics of Alintegimod monotherapy by measuring Area Under the Curve (AUC) | 1 year
  To characterize the pharmacokinetics of AUC of Alintegimod monotherapy.
Characterize Pharmacokinetics of Alintegimod plus ipilimumab by measuring Maximum Plasma Concentration (Cmax) | 1 year
  To characterize the pharmacokinetics of Cmax of Alintegimod in combination with ipilimumab.
Characterize Pharmacokinetics of Alintegimod plus ipilimumab by measuring Area Under the Curve (AUC) | 1 year
  To characterize the pharmacokinetics of AUC of Alintegimod in combination with ipilimumab.
Determine Progression Free Survival (PFS) response in patients treated with Alintegimod plus ipilimumab followed by nivolumab using RECIST v1.1 tumor assessment criteria. | 18 months
  To assess the progression-free survival of patients treated with Alintegimod in combination with ipilimumab followed by nivolumab monotherapy, using RECIST v1.1 assessment for progression.
Determine Overall Response Rate (ORR) in patients treated with Alintegimod plus ipilimumab followed by nivolumab using RECIST v1.1 response assessment criteria. | 18 months
  To assess the overall response rate of patients treated with Alintegimod in combination with ipilimumab followed by nivolumab monotherapy, using RECIST v1.1 assessment for progression.

CONTACTS AND LOCATIONS:
Overall Officials: Lionel Lewis, MA, MB.Bch, MD, Study Chair — 7 Hills Pharma
Locations (4):
- United States (4):
  - Florida Cancer Specialists, Lake Mary, Florida
  - Dartmouth Hitchcock, Lebanon, New Hampshire
  - Brown University Health Cancer Institute, Providence, Rhode Island
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided